CLINICAL TRIAL: NCT03912285
Title: Pharmacokinetic and Hemodynamic Interactions Between Amlodipine and Losartan in Humans
Brief Title: The Pharmacokinetic Interaction Between Amlodipine and Losartan
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Korea University Anam Hospital (Other)
Collaborators: Hanmi Pharmaceutical co., ltd. (Other)
Responsible Party: Principal Investigator, Ji-Young Park, Professor, Korea University Anam Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HM-ALOS-101
Record Dates: First submitted 2019-04-09; First posted 2019-04-11 (Actual); Last update posted 2019-04-12 (Actual); Status verified 2019-04

CONDITIONS: Healthy
MeSH Terms: interventions — Losartan; Amlodipine

STUDY DESIGN:
Intervention Model Description: an open-label, three-period, fixed-sequence clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Amlodipine, losartan, and amlodipine plus losartan (Experimental): Period 1:
  amlodipine 10mg will be administered orally once a day for 9 days.
  Period 2:
  losartan 100mg will be administered orally once a day for 9 days after 13 days of the washout period.
  Period 3:
  amlodipine 10mg once a day plus losartan 100mg once a day will be administered orally for 9 days after 6 days of the washout period.
  Interventions: Drug: Amlodipine10mg; Drug: Losartan potassium 100mg; Drug: Amlodipine plus Losartan

INTERVENTIONS:
Drug: Amlodipine10mg — Amlodipine 10mg will be administered orally twice a day for 9 days
Drug: Losartan potassium 100mg — Losartan 100mg will be administered orally once a day for 9 days
Drug: Amlodipine plus Losartan — Amlodipine plus Losartan same way as "arm: amlodipine" and "arm: losartan"

SUMMARY:
This clinical trial aims to assess the pharmacokinetic interaction between amlodipine and losartan in healthy male subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers aged between ≥ 20 and ≤ 45 years old
2. Weight ≥ 50kg, with calculated body mass index(BMI) of ≥ 18 and ≤ 29.9kg/m²
3. Subjects who agree to use a combination of effective contraceptive methods or medically acceptable contraceptive methods for up to 28 days after the date of administration of the clinical trial drug and agree not to provide sperm
4. Subject who are informed of the investigational nature of this study, voluntarily agree to participate in this study

Exclusion Criteria:

1. History or presence of a clinically significant and active cardiovascular, respiratory, hepatobiliary, renal, hematological, gastrointestinal, endocrine, immune, dermatologic, neurologic or psychiatric disorder
2. With symptoms indicating acute illness within 28 days prior to the first Investigational Product administration
3. Any medical history that may affect drug absorption, distribution, metabolism, and excretion
4. Genetic problems such as galactose intolerance, Lapp lactose dehydrogenase deficiency or glucose-galactose uptake disorder
5. Any clinically significant active chronic disease

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01-10 (Actual); Primary Completion 2009-03-17 (Actual); Study Completion 2009-06-09 (Actual)

PRIMARY OUTCOMES:
AUCtau(area under the plasma concentration-time curve for a dosing interval at steady state) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46
Cmax,ss(Maximum plasma concentration of the drug at steady state) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46

SECONDARY OUTCOMES:
Cmin,ss(Minimum concentration of the drug in plasma at steady state) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46
Tmax,ss(Time to maximum plasma concentration at steady state) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46
1/2(Terminal elimination half-life) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46
CLss/F(Apparent total body clearance of the drug from plasma at steady state) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46
Vd,ss/F(Apparent volume of distribution at steady state) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46
PTF(Peak-to-trough fluctuation) | 0 (predose) ~ 24 hours at day 9, day 31, and day 46

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Clinical Pharmacology & Toxicology, Anam Hospital, Korea University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No